CLINICAL TRIAL: NCT02956538
Title: Induced Adult Refractory Active Crohn's Disease Clinical Relieving by Using Thalidomide: A Randomized, Double-blind, Placebo-controlled Multicenter Clinical Study
Brief Title: Induced Adult Refractory Active Crohn's Disease Clinical Relieving by Using Thalidomide
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiang Gao, Clinical Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2016022
Record Dates: First submitted 2016-10-13; First posted 2016-11-07 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Thalidomide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- thalidomide (Experimental): thalidomide 100mg tablet by mouth, every night for 8 weeks
  Interventions: Drug: Thalidomide
- placebo (Active Comparator): placebo (for thalidomide) 100mg tablet by mouth, every night for 8 weeks
  Interventions: Drug: placebo(for thalidomide)

INTERVENTIONS:
Drug: Thalidomide
  Arms: thalidomide
Drug: placebo(for thalidomide) — sugar pill manufactured to mimic thalidomide 100mg tablet
  Arms: placebo

SUMMARY:
With the development and application of biological agents, the treatment effect was considerable degree improvement on refractory corn's disease. However, there are quite a part of the CD patients lost response during treatment of using response. Moreover, due to various reasons, there still a lot limited on the using of biological agents in China, that make quite a part of the refractory CD patients lack of further medical treatment options. There has been a RCT study which prove that thalidomide effect and safety on treating refractory CD or who were lost response by using biological agents in Italy, but the object of study is only limited in children and adolescents. There are some small sample studies also confirmed the efficacy and safety on refractory corn's disease by using thalidomide, but need more RCT evidence.

DETAILED DESCRIPTION:
It will be divided two groups of patients by using randomized, double-blind. One group was treated by thalidomide, the other was placebo. It will be unlocked blind and analysis the effect and safety about thalidomide after 8 weeks. The second, patients still use thalidomide after unlock blind to prove its longtime treatment effect and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years old
* Diagnosis of patients with CD
* Disease in the activity: CDA Ⅰ > 150 points, endoscopic see active lesions
* Refractory: immunosuppressive drugs or biological agents which are used in current treatment is invalid and/or intolerance

Exclusion Criteria:

* Fiber stenosis caused by gastrointestinal obstruction symptoms
* Fistula exclude anal fistula
* Pregnancy or lactation
* Period of women have fertility program during the study
* Treatment not foot eight weeks after last IFX
* Central or peripheral nerve disease
* Abnormal in liver and renal function
* Heart function failure
* Malignant tumor
* Active tuberculosis

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
difference CDAI between thalidomide group and placebo group | 8 weeks
  CDAI means Crohn's Disease Activity Index.The purpose of this crohn's disease activity index (CDAI) calculator is to gauge the progress or lack of progress for people with crohn's disease. The reference article says "generally speaking, CDAI scores below 150 indicate a better prognosis than higher scores."
difference SES-CD score between thalidomide group and placebo group | 8weeks
  SES-CD means Simple endoscopic score for Crohn's disease ,which predicts long-term prognosis in Crohn's disease patients with clinical remission.

SECONDARY OUTCOMES:
difference CDAI between different thalidomide dosage group | 1 year
  CDAI means Crohn's Disease Activity Index.The purpose of this crohn's disease activity index (CDAI) calculator is to gauge the progress or lack of progress for people with crohn's disease. The reference article says "generally speaking, CDAI scores below 150 indicate a better prognosis than higher scores."
difference SES-CD score between different thalidomide dosage group | 1 year
  SES-CD means Simple endoscopic score for Crohn's disease ,which predicts long-term prognosis in Crohn's disease patients with clinical remission.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang gao, MD, Study Chair — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Department of Gastroenterology, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes